CLINICAL TRIAL: NCT00301327
Title: A Multi-Center, Randomized, Vehicle Controlled, Double Blind Clinical Trial to Evaluate the Efficacy and Safety of Summers Non-Pesticide Lice Asphyxiator (L.A.) for the Treatment of Head Lice.
Brief Title: Efficacy and Safety of Summers Non-Pesticide Lice Asphyxiator (L.A.)for the Treatment of Head Lice.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Summers Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SU-01-2005
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Head Lice

INTERVENTIONS:
Drug: Summers 5% L.A.

SUMMARY:
This is a multi-center, randomized, double blind, vehicle controlled, study designed to evaluate the pediculicidal activity of Summers 5% L.A. compared to a vehicle control.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 6 months of age or older.
2. Have an active infestation with pediculus capitis, the human head louse, with at least three live lice at baseline.
3. Agree not to use any other pediculicides or medicated hair-grooming products during the duration of the study.
4. Be healthy, non-febrile, and not suffering from an infection likely to require antibiotic therapy during the study period.
5. Subject or guardian is able to understand the new HIPAA regulations and sign the HIPAA form.
6. Subject or guardian has read, understood, and signed appropriate informed consent in English. If English is not the primary language, the information about the study must be explained in their language and a copy of the informed consent must be in that language.
7. Subject is willing to participate in the study, and abide by the protocol requirements.

   -

Exclusion Criteria:

1. Participation in any clinical study within the past 30 days.
2. Known hypersensitivity to any ingredient in the product formulation.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2006-01

PRIMARY OUTCOMES:
Treatment success is defined as the absence of live lice.

SECONDARY OUTCOMES:
The cumulative proportions of subjects determined to be treatment failures at the Second Evaluation Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Meinking, Principal Investigator — Global Health Associates of Miami; Anne Lucky, Dr., Principal Investigator — Dermatology Research Associates; Jon Thomas, Dr., Principal Investigator — Alegent Health; E.A. Clark, Dr., Principal Investigator — Diagnostic Clinic of Longview, TX; Peter E Silas, Dr., Principal Investigator — Advanced Clinical Research Institute
Locations (5):
- United States (5):
  - Global Health Associates of Miami 7800, SW 57 Avenue, Suite 219E, Miami, Florida
  - Alegent Health, Harmony Street, 2nd Floor, Council Bluffs, Iowa
  - Dermatology Research Associates 7691 Five Mile Road, Suite 312, Cincinnati, Ohio
  - Diagnostic Clinic of Longview, TX 707 Hollybrook Drive, Longview, Texas
  - Wee Care Pediatrics, 1580 West Antelope Drive, Suite 100, Layton, Utah

REFERENCES:
- [Derived] Meinking TL, Villar ME, Vicaria M, Eyerdam DH, Paquet D, Mertz-Rivera K, Rivera HF, Hiriart J, Reyna S. The clinical trials supporting benzyl alcohol lotion 5% (Ulesfia): a safe and effective topical treatment for head lice (pediculosis humanus capitis). Pediatr Dermatol. 2010 Jan-Feb;27(1):19-24. doi: 10.1111/j.1525-1470.2009.01059.x. PMID 20199404
- See also: Related Info — http://www.sumlab.com